CLINICAL TRIAL: NCT05539456
Title: Reliability and Validity of the Turkish Version of the PedsQL 3.0 Neuromuscular Module for 2-to 4- Year-old: a Quality-of-life Measure for Patients With Spinal Muscular Atrophy in Turkey
Brief Title: Reliability and Validity of the Turkish Version of the PedsQL 3.0 Neuromuscular Module for 2-to 4- Year-old
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-772.02-213
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Spinal Muscular Atrophy; Quality of Life; Neuromuscular Diseases; Pediatric Disorder
Keywords: Spinal Muscular Atrophy; Quality of Life; Neuromuscular Diseases
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the investigator's study was to investigate translating the PedsQL 3.0 Neuromuscular Module for 2-to 4- Year-old and using it in clinics reliably and validity with a Turkish version of the PedsQL Generic Core (Pediatric Quality of Life Questionnare) in children with Spinal Muscular Atrophy in Turkey

DETAILED DESCRIPTION:
The PedsQL 3.0 Neuromuscular Module for 2-to 4- year-old will be translated into Turkish by following the language translation steps. First of all, the English form will be translated into Turkish by two people who are fluent in English. Then, the forms translated by another expert in the field will be reviewed. The revised text will be translated from Turkish into English by another person with a good command of English and will be compared with the original scale by the lecturer. If a significant change in meaning is not detected, the scale will be applied to 10 parents. In case of incomprehensible questions, which are reported to be lacking in expression, the scale will be finalized after revision and corrections are made by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with spinal muscular atrophy
* Having a child between the ages of 2-4
* Accept to participate in the study

Exclusion Criteria:

* Lack of cooperation during work
* Presence of disease other than SMA, which will prevent participation in the study

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spinal muscular atrophy between 2 to 4 years age.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
PedsQLTM 3.0 neuromuscular module for 2-to 4- Year-old | 5-10 minutes
  The module encompasses three scales:
  1. About My/My Child's Neuromuscular Disease (17 items),
  2. Communication (3 items),
  3. About Our Family Resources (5 items).
  The scale is comprised a parent proxy-report format for children ages 2 to 4 years.
  Items in all forms are essentially identical but contain slightly different language for first or third person tense.
  The participants are asked how much of a problem each item had been during the past month.
  Responses are rated on a 5-point Likert scale across child self-report for children, teens, and parent proxy-reports (0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem, 4 = almost always a problem).
  Items are linearly transformed to a 0 to 100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0) so that higher scores indicate better HRQOL.

SECONDARY OUTCOMES:
PedsQLTM 4.0 generic core scales | 5-10 minutes
  The 23-item PedsQLTM 4.0 Generic Core Scales encompass:
  1. Physical Functioning (8 items),
  2. Emotional Functioning (5 items),
  3. Social Functioning (5 items),
  4. School Functioning (5 items)
  The formats, instructions, Likert scales, and scoring methods are the same as those of the PedsQLTM 3.0 Neuromuscular Module. To create the Psychosocial Health Summary Score, the mean is computed as the sum of the items divided by the number of items answered in the Emotional, Social, and School Functioning Subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Kutlutürk Yıkılmaz, Principal Investigator — Medipol University
Locations (1):
- Seval Kutlutürk Yıkılmaz, Istanbul, Kavacık, Turkey (Türkiye)